CLINICAL TRIAL: NCT03112902
Title: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Compelling insights impacting the scientific rationale
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 16-1875
Record Dates: First submitted 2017-03-24; First posted 2017-04-13 (Actual); Results first posted 2021-07-21 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (10):
- Effects of tACS during SWS- Standard/Nested 1 (Active Comparator): This is a triple cross-over with a sham control condition; the standard tACS administered first, then Nested, then sham.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Older Adults Active 1 (Active Comparator): This is a double cross-over with a sham control condition; the tACS administered first, then the sham
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- MCI Active 1 (Active Comparator): This is a cross-over with a sham control condition; the standard tACS administered first, then sham.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Standard/Nested 2 (Active Comparator): This is a triple cross-over with a sham control condition; the standard tACS administered first, then sham, then nested tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Standard/Nested 3 (Active Comparator): This is a triple cross-over with a sham control condition; the sham tACS administered first, then nested tACS, then standard tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Older Adults Active 2 (Active Comparator): This is a double cross-over with a sham control condition; the sham administered first, then the tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- MCI Active 2 (Active Comparator): This is a cross-over with a sham control condition; the sham administered first, then standard tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Standard/Nested 4 (Active Comparator): This is a triple cross-over with a sham control condition; the sham tACS administered first, then standard tACS, then nested tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Standard/Nested 5 (Active Comparator): This is a triple cross-over with a sham control condition; the nested tACS administered first, then sham, then standard tACS.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance
- Effects of tACS during SWS- Standard/Nested 6 (Active Comparator): This is a triple cross-over with a sham control condition; the nested tACS administered first, then standard tACS, then sham.
  Interventions: Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance

INTERVENTIONS:
Device: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance — Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.

SUMMARY:
Loss of slow wave sleep (SWS) is common in mild cognitive impairment (MCI) and Alzheimer's disease, and is thought to worsen thinking, memory and brain degeneration. Initial studies suggest that correction of sleep deterioration may slow the progression of brain damage in mild cognitive impairment, and might be able to stop the development of Alzheimer's disease. Transcranial alternating current stimulation (tACS) uses electrodes to deliver very small amounts of electricity through the brain, with direct effects on brain cell function. Transcranial electric stimulation has been demonstrated to enhance slow wave sleep and to improve memory when applied during sleep in healthy adults. The purpose of this research is to investigate tACS to modulate sleep, thinking/memory, mood, and quality of life among normal healthy adults, older adults, as well as individuals with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-85
* Native English speakers
* Neurological diagnosis of amnestic mild cognitive impairment (aMCI)

Exclusion Criteria:

* brain tumors
* skull defects
* epilepsy
* metal implants/devices above the neck
* eczema or sensitive skin
* insomnia
* sleep apnea that requires use of a CPAP machine
* rapid eye movement (REM)-sleep behavior disorder
* currently pregnant or trying to become pregnant during the study period
* diagnosis of cognitive impairment *cognitive impairment required for MCI arms

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2021-05-04 (Actual); Study Completion 2021-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brice McConnell, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado AMC, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Effects of tACS During SWS- Standard/Nested 1: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This is a triple crossover study design: standard tACS first, then nested tACS, then sham.
- Effects of tACS During SWS- Standard/Nested 2: This is a triple crossover study design: standard tACS first, then sham, then nested tACS.
- Effects of tACS During SWS- Standard/Nested 3: This is a triple crossover study design: sham first, then nested tACS, then standard tACS.
- Effects of tACS During SWS- Standard/Nested 4: This is a triple crossover study design: sham first, then standard tACS, then nested tACS.
- Effects of tACS During SWS- Standard/Nested 5: This is a triple crossover study design: nested tACS first, then sham, then standard tACS.
- Effects of tACS During SWS- Standard/Nested 6: This is a triple crossover study design: nested tACS first, then standard tACS, then sham.
- Effects of tACS During SWS- Older Adults Active 1; Effects of tACS During SWS- MCI Active 1: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This is a crossover study design: standard tACS first, then sham.
- Effects of tACS During SWS- Older Adults Active 2; Effects of tACS During SWS- MCI Active 2: This is a crossover study design: sham first, then standard tACS.
Period: Overall Study
Arm/Group | Effects of tACS During SWS- Standard/Nested 1 | Effects of tACS During SWS- Standard/Nested 2 | Effects of tACS During SWS- Standard/Nested 3 | Effects of tACS During SWS- Standard/Nested 4 | Effects of tACS During SWS- Standard/Nested 5 | Effects of tACS During SWS- Standard/Nested 6 | Effects of tACS During SWS- Older Adults Active 1 | Effects of tACS During SWS- Older Adults Active 2 | Effects of tACS During SWS- MCI Active 1 | Effects of tACS During SWS- MCI Active 2
Started | 2 | 2 | 3 | 1 | 1 | 3 | 9 | 3 | 0 | 0
Completed | 0 | 2 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not Completed | 2 | 0 | 1 | 1 | 0 | 3 | 8 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated prior to completion enrollment, and prior to any enrollment of MCI arm.
Groups:
- Effects of tACS During SWS- Standard/Nested 1: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This is a triple crossover: standard tACS, then nested tACS, then sham.
- Effects of tACS During SWS- Standard/Nested 2; Effects of tACS During SWS- Standard/Nested 6: This is a triple crossover: nested tACS, then standard tACS, then sham.
- Effects of tACS During SWS- Standard/Nested 3: This is a triple crossover: sham, then nested tACS, then standard tACS.
- Effects of tACS During SWS- Standard/Nested 4: This is a triple crossover: sham, then standard tACS, then nested tACS
- Effects of tACS During SWS- Standard/Nested 5: This is a triple crossover: nested tACS, then sham, then standard tACS
- Effects of tACS During SWS- Older Adults Active 1; Effects of tACS During SWS- MCI Active 1: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This is a crossover: standard tACS, then sham.
- Effects of tACS During SWS- Older Adults Active 2; Effects of tACS During SWS- MCI Active 2: This is a crossover: sham, then tACS.
- Total: Total of all reporting groups
Arm/Group | Effects of tACS During SWS- Standard/Nested 1 | Effects of tACS During SWS- Standard/Nested 2 | Effects of tACS During SWS- Standard/Nested 3 | Effects of tACS During SWS- Standard/Nested 4 | Effects of tACS During SWS- Standard/Nested 5 | Effects of tACS During SWS- Standard/Nested 6 | Effects of tACS During SWS- Older Adults Active 1 | Effects of tACS During SWS- Older Adults Active 2 | Effects of tACS During SWS- MCI Active 1 | Effects of tACS During SWS- MCI Active 2 | Total
Number analyzed (Participants) | 2 | 2 | 3 | 1 | 1 | 3 | 9 | 3 | 0 | 0 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 3 | 1 | 1 | 3 | 4 | 1 | 0 | 0 | 17
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 0 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 1 | 2 | 4 | 2 | 0 | 0 | 12
  Male | 0 | 2 | 3 | 0 | 0 | 1 | 5 | 1 | 0 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 3 | 1 | 1 | 2 | 9 | 3 | 0 | 0 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  White | 2 | 2 | 3 | 1 | 1 | 3 | 8 | 2 | 0 | 0 | 22
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 3 | 1 | 1 | 3 | 9 | 3 |  |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Electro-encephalogram (EEG) Power of Slow Wave Oscillations
Description: Power of EEG data in microvolts within slow wave frequency range.
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Groups:
- Effects of tACS During SWS- Standard: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This was part of a triple crossover
- Effects of tACS During SWS- Nested: This was part of a triple crossover
- Effects of tACS During SWS- Older Adults Active; Effects of tACS During SWS- MCI Active: This is a cross-over with a sham control condition
  Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Change in Declarative Memory Encoding
Description: Word-paired associations
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject.
Population: Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for the study outcome measures.
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Change in Procedural Memory Encoding *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Finger tapping task *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Change in Sleep Architecture as Measured by Minutes in Each Stage of Sleep *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: EEG data *No processing of data occurred to provide information about this outcome measure.
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Change in Fast and Slow Spindle Numbers During Sleep *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: EEG data *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Change in Slow Wave Coherence *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: as for outcome 5
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Change in Slow Wave Power *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: as for outcome 5
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Change in Sleep Architecture as Measured by Self Reported Sleep Timing *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Sleep diary for subjective experience *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change in Hospital Anxiety and Depression Scale (HADS) *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Mood outcome *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Change in Clinical Global Impression of Change (CGIC) *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Global assessment *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Change in Battery of Working Memory Tasks *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Assessment of working memory *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change in Battery of Attention Tasks *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Assessment of attention *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change in Battery of Visuospatial Processing Tasks *No Processing of Data Occurred to Provide Information About This Outcome Measure.
Description: Assessment of visuospatial ability *Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed. No data was analyzed for this outcome measure
Time Frame: Before and after each night of study session, up to 24 weeks from enrollment for each subject
Population: as for outcome 2
Arm/Group | Effects of tACS During SWS- Standard | Effects of tACS During SWS- Nested | Effects of tACS During SWS- Older Adults Active | Effects of tACS During SWS- MCI Active
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 months (approx)
Description: Adverse events were monitored after every period of participant data collection/study visit.
Groups:
- Effects of tACS During SWS- Standard/Nested 1: Application of Transcranial Alternating Current Stimulation for Modulation of Sleep and Cognitive Performance: Transcranial Alternating Current Stimulation will be applied during slow wave sleep to assess effects on memory and sleep architecture.
  This is a triple crossover: standard tACS, then nested, then sham
- Effects of tACS During SWS- Standard/Nested 2: This is a triple crossover: standard tACS, then sham, then nested tACS
- Effects of tACS During SWS- Standard/Nested 3: This is a triple crossover: sham, then nested tACS, then standard tACS,
- Effects of tACS During SWS- Standard/Nested 4: This is a triple crossover: sham, then standard tACS, then nested tACS,
- Effects of tACS During SWS- Standard/Nested 5: This is a triple crossover: nested tACS, then sham, then standard tACS,
- Effects of tACS During SWS- Standard/Nested 6: This is a triple crossover: nested tACS, then standard tACS then sham.
- Effects of tACS During SWS- Older Adults Active 2; Effects of tACS During SWS- MCI Active 2: This is a crossover: sham and then standard tACS
Arm/Group | Effects of tACS During SWS- Standard/Nested 1 | Effects of tACS During SWS- Standard/Nested 2 | Effects of tACS During SWS- Standard/Nested 3 | Effects of tACS During SWS- Standard/Nested 4 | Effects of tACS During SWS- Standard/Nested 5 | Effects of tACS During SWS- Standard/Nested 6 | Effects of tACS During SWS- Older Adults Active 1 | Effects of tACS During SWS- Older Adults Active 2 | Effects of tACS During SWS- MCI Active 1 | Effects of tACS During SWS- MCI Active 2
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/1 | 0/1 | 0/3 | 0/9 | 0/1 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/1 | 0/1 | 0/3 | 0/9 | 0/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/3 | 0/1 | 0/1 | 0/3 | 0/9 | 0/3 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
During this trial we made compelling discoveries into the nature of slow wave sleep that undermined the rationale and data analysis plan for this trial. Problems and new insights related to the study's design were encountered during data collection that fundamentally affected the rationale and feasibility of the trial. Trial was terminated before sufficient data could be collected and analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/02/NCT03112902/Prot_002.pdf
  • Statistical Analysis Plan (2021-06-06): https://cdn.clinicaltrials.gov/large-docs/02/NCT03112902/SAP_003.pdf